CLINICAL TRIAL: NCT03026803
Title: A Phase II Study of Oxaliplatin and Capecitabine in Unresectable Metastatic Hepatocellular Cancer
Brief Title: A Study of Oxaliplatin and Capecitabine in Unresectable Metastatic Hepatocellular Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Sorafenib became first line treatment for HCC, the designed treatment became less competitive. The company Sanofi decided not to continue to support
Sponsor: City of Hope Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05195
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Liver Cancer; Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin and Capecitabine (Experimental): 21 day cycle with Oxaliplatin 50mg/m2 day 1 and day 8 administered IV, Capecitabine 750 mg/m2 bid p.o. daily from day 1 to day 14
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
  Other Names: Eloxatin
Drug: Capecitabine — Given PO
  Other Names: Xeloda

SUMMARY:
This phase II trial is studying how well giving oxaliplatin and capecitabine together works in treating patients with liver cancer.

DETAILED DESCRIPTION:
Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving these drugs together may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed hepatocellular carcinoma which is recurrent, metastatic or unresectable.
* Patients may have up to two prior chemotherapy regimes. In addition, they may have had previous radiation, chemoembolization, and/or alcohol injections.
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, and which has clearly progressed during the observation interval prior to participation in this study. Pleural effusions and ascites will not be considered measurable, but may be present in addition to the measurable lesion(s).
* Karnofsky performance status > 70%.
* Patients should have an expected survival of at least 2 months.
* Leukocytes >3,000/µl
* Absolute neutrophil count >1,500/µl
* Platelets >50,000/µl
* Total bilirubin < 3.0 g/dl
* AST (aspartate aminotransferase) (serum glutamic oxaloacetic transaminase(SGOT)/ALT (alanine aminotransferase) (serum glutamic pyruvic transaminase)(SGPT) < 5 times institutional upper limit of normal
* Creatinine < 2.0 OR measured or calculated creatinine clearance >60 mL/min for patients with creatinine levels above institutional normal
* Brain metastasis is not an exclusion, however, patients are only eligible if they have had successful control of the brain tumor(s) by surgery or stereotactic RT.
* Patients with no evidence of clinically significant neuropathy.
* All prior therapy must have been completed at least 4 weeks prior to the patient's entry on this trial.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Breastfeeding should be discontinued if the mother is treated with oxaliplatin.
* Subjects with chronic hepatitis B or C may be undergoing treatment with α interferon and/or ribavirin, as long as they meet the other criteria for entry on to this study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients have prior oxaliplatin or xeloda treatment or undergoing therapy with other investigational agents.
* History of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia.
* HIV-positive patients receiving anti-retroviral therapy (HAART) are excluded from the study because of possible pharmacokinetic interactions.
* Patients with a diagnosis of pulmonary fibrosis or a pulmonary interstitial process.
* Patients unable to swallow capecitabine will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yen, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaliplatin and Capecitabine: 21 day cycle with Oxaliplatin 50mg/m^2 day 1 and day 8 administered IV, Capecitabine 750 mg/m^2 bid p.o. daily from day 1 to day 14
  Oxaliplatin: Given IV
  Capecitabine: Given PO
Period: Overall Study
Arm/Group | Oxaliplatin and Capecitabine
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin and Capecitabine
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 71 [65 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Oxaliplatin and Capecitabine
Number analyzed (Participants) | 4
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Oxaliplatin and Capecitabine
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin and Capecitabine (N=4)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin and Capecitabine (N=4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Creatinine increased (Investigations) | 2 (3)
Leukocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (4)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (6)
Taste alteration (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (5)
Flushing (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to Sorafenib becoming a first line treatment for HCC, the designed treatment became less competitive. The company Sanofi decided not to continue support. Study was terminated after accrual of 4 of the 32 planned patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes